CLINICAL TRIAL: NCT05384704
Title: Evaluating the Effectiveness of Empower@Home for Depression Among Older Adults
Brief Title: A Single Group Study of Empower@Home-an Internet Cognitive Behavioral Therapy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Xiaoling Xiang, Xiaoling Xiang, PhD, MSW, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00212950
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders
Keywords: Cognitive Behavioral Therapy; Older Adults; Internet-Based Intervention; Depression; Social Isolation
MeSH Terms: conditions — Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders; Social Isolation

STUDY DESIGN:
Intervention Model Description: The purpose of this research project is to assess the effectiveness of a novel internet-based cognitive behavioral therapy (iCBT) program called Empower@Home. The program is intended to decrease depression in participants by encouraging them to participate in meaningful and enjoyable activities while challenging problematic thinking patterns.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-based program (Experimental): Participants will be provided with access to a 9-session online program and will receive supportive remote assistance throughout regarding technical and programmatic issues.
  Interventions: Behavioral: Empower@Home

INTERVENTIONS:
Behavioral: Empower@Home — The intervention is a 9-week course of internet-based cognitive behavioral therapy. During the active intervention phase, participants will receive weekly support from a trained research staff.

SUMMARY:
This is a single group study of a novel internet-based cognitive behavioral therapy program for older adults with elevated depressive symptoms. This study will enroll approximately 300 older adults throughout the state of Michigan to test the effectiveness of Empower@Home with older adults. The intervention will take approximately 10 weeks to complete. Participants will have lower levels of depression after completing the intervention than before enrollment. Participants will be able to use the internet-based platform with minimal support.

DETAILED DESCRIPTION:
Depression affects up to 40% of homebound seniors but most homebound seniors do not receive psychotherapy due to various access barriers. The study team focuses on developing community-based solutions to reduce these access barriers. In a previously approved project HUM00207612, the study team tested the feasibility of a novel internet-based cognitive behavioral therapy (iCBT) program called Empower@Home. The pilot project allowed refining study procedures and the web platform used to deliver the program. In this new project, the study team will conduct a larger single group study to test the effectiveness of Empower@Home with older adults. Recruitment methods include 1) referrals from social service agencies and 2) advertisements on social media and the program website.

The intervention involves attending up to 9 pre-recorded online therapy sessions and receiving weekly coaching calls from trained research assistants for up to 10 weeks. Participants will engage in therapy in their private homes. Three assessments are scheduled, including a comprehensive baseline, a post-test, and a 10-week follow-up. Each assessment takes about 40 minutes to complete over the phone or via an online survey, depending on the participants' preference.

Subjects will be recruited from agency referrals and advertisements. Between May 2022 and Dec 2023, about 300 subjects will be recruited into a single group study design where all eligible and consented participants will receive the intervention immediately without waiting.

ELIGIBILITY:
Inclusion Criteria:

1. ≥50 years
2. have at least mild depressive symptoms, based on PHQ-9 >=5
3. are willing to participate

Exclusion Criteria:

1. Probable cognitive impairment based on the Blessed Orientation, Memory, and Concentration scale (score >9).
2. They do not speak English
3. have active suicidal ideation, defined as moderate to high risk based on the 6-item Columbia-Suicide Severity Rating Scale (C-SSRS)
4. Have a terminal illness or unstable physical health with a high risk of hospitalization within the next 3 months
5. Have severe vision impairment that can not be corrected and with no in-home help to assist them with using a mobile device
6. possible substance use disorders as assessed by the 4-item CAGE screener (>=2 on the CAGE AND have not been sober for at least one year)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Change from Baseline PHQ-9 at 10 weeks
  Change in 9 item standardized measures of depressive symptom severity. PHQ-9 score ranges from 0 to 27, with a higher score indicating more severe symptoms.
Modified Treatment Evaluation Inventory | 10 weeks
  11-item Likert scale relating to acceptability of program to participant modified for older adults and the study context. The score ranges from 11 to 55, and a higher score means higher acceptability.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder Assessment-7 (GAD-7) | Change from Baseline at 10 weeks
  Change in 7-item standardized measure for severity of anxiety symptoms. GAD7 score ranges from 0 to 21, higher score means more severe symptoms.
Change in Duke Social Support Index (DSSI)-10 | Change from Baseline at 10 weeks
  Change in 10 item standardized measure for social interaction and satisfaction with social support. Total score ranges from 10 to 30, higher score means higher social support.
Change in PROMISE-SI | Change from Baseline at 10 weeks
  Change in 8 item standardized measure for feelings of loneliness. Total score ranges from 8 to 40, higher score means higher levels of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Xiang, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT05384704/ICF_000.pdf